CLINICAL TRIAL: NCT03282214
Title: A Self-Management Energy Conservation Program for Cancer-Related Fatigue in Thai Women With Breast Cancer Receiving Chemotherapy: A Pilot Study
Brief Title: A Self-Management Energy Conservation Program for Cancer-Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Wipasiri Naraphong, Postdoctoral Fellow, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D43TW009883 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Cancer-related Problem/Condition; Cancer, Breast; Fatigue
Keywords: Energy conservation; Self management
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management energy conservation (Experimental): Thai women with breast cancer randomized to the group will receive four sessions approximately every three weeks with the PI. The women will be instructed on how to do a self-management energy conservation program.
  Interventions: Behavioral: Self-management energy conservation
- Control (No Intervention): The participants will be given two pamphlets (general issues about breast cancer and self-care activities for patients receiving chemotherapy) provided by the health care team at the study sites. The participants in the control group will be encouraged to maintain their current daily activities during the 12-week period The participants will wear a pedometer to record the number of steps which is one of the activity outcomes.

INTERVENTIONS:
Behavioral: Self-management energy conservation — The experimental group will receive four sessions approximately every three weeks with the PI. These sessions will correspond to the cycles of chemotherapy they will receive, with the first two sessions being during cycle 1, and sessions 3 and 4 being during cycles 2 and 3 of chemotherapy, respectively. The women will be instructed on how to assess their activity patterns by making a list prioritizing their usual activities. The journal and priority list (a "to do" list) provide the basis for the second session. In this session, the participant will learn to create a plan for managing valued activities to minimize the amount of energy used, to report the fatigue experienced during and after an activity done in the journal and will learn strategies to manage fatigue and optimize activity. In the third session, the participant will evaluate and revise their individualized plan. In addition, the participant will be instructed to wear a pedometer to record objective physical activity.
  Arms: Self-management energy conservation

SUMMARY:
The purpose of this pilot study is to examine a 12-week self-management energy conservation program (ECAM)'s effects on fatigue, and secondarily on sleep, physical activity, anxiety and depression, self-efficacy, and beliefs about fatigue in a group of Thai women with breast cancer who are undergoing chemotherapy. We will also evaluate how well women like the intervention, how easy it is to use and whether women will do the activities.

DETAILED DESCRIPTION:
Cancer-related fatigue is a distressing and multidimensional symptom. Research in the US has explored the efficacy of energy conservation interventions for fatigue and related symptoms but no previous ECAM programs have been tested in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Thai women are age 18 or older; are diagnosed with stage I-III breast cancer; are scheduled to receive at least four cycles of chemotherapy given in 21-day-intervals; report at least 4 out of 10 or higher on a fatigue scale in the past month; are able to read and write in Thai and can be contacted by telephone.

Exclusion Criteria:

* Thai women have a history of severe psychiatric illness, or have other illnesses that could be responsible for the fatigue other than cancer such as iron deficiency anemia, multiple sclerosis, congestive heart failure, chronic fatigue syndrome or fibromyalgia. With regard to anemia, women must have a certain hemoglobin in the normal range at baseline. They also cannot have acute or chronic bone, joint, or muscular abnormalities that would increase the risk of falls and injury. Women scheduled to receive concurrent radiation therapy are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Thai women
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue (CRF) | Change from baseline CRF scores at 12 weeks
  A 22-item scale, 0 to 10 numerical scaling, with four dimensions of fatigue will be used to measure CRF severity.

SECONDARY OUTCOMES:
Acceptability | at 12 weeks
  Open-ended questions will be used to ask about the most positive and negative aspects of the intervention, what modules did they use the most, what were barriers to using the intervention, what would they like to see added or deleted in future modules, and any suggestions on how the program could be improved.
Satisfaction | at 12 weeks
  Scaling questions about satisfaction with the intervention will be responded on a 5-point scale (1 = dissatisfied to 5 = completely satisfied).
The General Sleep Disturbance (GSD) | Change from baseline GSD scores at 12 weeks
  A 21-item, eight-point Likert scale from 0 (never) to 7 (every day) will be used to measure subjective sleep disturbance.
Physical Activity (subjective measure) | Change from baseline GSLTPAG scores at 12 weeks
  Godin Leisure-Time Physical Activity Questionnaire (GSLTPAQ): A 4-item self-administered questionnaire asking information about the number of times one engages in mild, moderate, and strenuous leisure-time physical activity bouts of at least 15 minutes duration in a week, and also asking how often participants typically engage in any regular activity until sweating or a racing heart on a scale of often, sometimes, never or rarely.
Physical Activity (objective measure) | Changes from baseline steps per day at 12 weeks
  A pedometer will be used to assess how many steps are taken each day.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS scores at 12 weeks
  The HADS is a 14-item questionnaire
Self-Efficacy for Managing Chronic Disease Scale (SEMCDS) | Change from baseline SEMCDS scores at 12 weeks
  This 6-item scale contain items will be used to measures self-reported current level of confidence to manage control the patient's symptoms, role function, emotional functioning, and communicating with physicians.
Fatigue Belief Questions (FBQ) | Change from baseline FBQ scores at 12 weeks
  A 20-item, six-point Likert scale from 1 (strongly disagree) to 6 (strongly agree) will be used to measure the fatigue beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: School of Nursing, Study Chair — University of Michigan
Locations (2):
- Thailand (2):
  - Saraburi Hospital, Changwat Sara Buri
  - Lopburi Cancer Hospital, Lopburi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion.

REFERENCES:
- [Derived] Naraphong W, Barton D. Self-Management Energy Conservation for Cancer-Related Fatigue in Thai Women With Breast Cancer Receiving Chemotherapy: A Pilot Study. Oncol Nurs Forum. 2023 Apr 21;50(3):337-347. doi: 10.1188/23.ONF.337-347. PMID 37155976